CLINICAL TRIAL: NCT00579384
Title: A Study of the Effects of JNJ-26489112 on the Photic Induced Paroxysmal Electroencephalogram Response in Patients With Photosensitive Epilepsy
Brief Title: A Study of the Effects of JNJ-26489112 on the Photic Induced Paroxysmal Electroencephalogram (EEG) Response in Patients With Photosensitive Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Associate Director, Experimental Medicine, Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CR014110; 26489112NAP2001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Photosensitive Epilepsy
Keywords: Photosensitive epilepsy; Reflex epilepsy; Epilepsy; JNJ-26489112
MeSH Terms: conditions — Epilepsy, Reflex; Epilepsy | interventions — N-((6-chloro-2,3-dihydrobenzo(1,4)dioxin-2-yl)methyl)sulfamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental)
  Interventions: Drug: JNJ-26489112; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-26489112 — Single oral dose of JNJ-26489112 up to 3000 mg on Day 2.
Drug: Placebo — Single dose of placebo on Day 1, and a second single dose of placebo on Day 3.

SUMMARY:
The purpose of this study is to check the Effects of JNJ-26489112 on the Photic Induced Paroxysmal electroencephalogram (EEG) Response in Patients with Photosensitive Epilepsy.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized (participants are assigned deliberately), single-blind (patients do not know which treatment they are receiving), within patient placebo-controlled study. Up to 32 male or female patients will participate in this study. The duration of subject participation is approximately 6 weeks.

Patients will receive the oral doses of study drug in the mornings of Days 1, 2, and 3. All patients will receive a single dose of placebo on Day 1, a single dose of JNJ-26489112 on Day 2, and a second single dose of placebo on Day 3. Blood samples will be taken for evaluation of JNJ-26489112 drug concentrations in plasma and blood. Blood samples will also be collected for laboratory safety assessments and measurement of antiepileptic drug concentrations. Further safety will be assessed by the reporting of adverse events, vital signs, 12-lead ECG, physical and neurological examinations. Patients will be discharged on the evening of Day 3 after the pharmacokinetic samples have been collected, and after assessment by the investigator, unless there are any ongoing adverse events which require in-house monitoring. EEG tracings, recorded during intermittent photic stimulation sessions, will be digitally recorded on a CD-ROM, coded and evaluated independently by one blinded clinical expert to determine the effects on the photosensitivity range. If complete suppression of photosensitivity or reduction of the photosensitivity range by at least 3 points on the photosensitivity scale in at least one eye condition (during closure, closed, open) is not observed in at least 3 of the 4 patients and a maximum tolerated dose has been reached, the study will be stopped. If reduction of the photosensitivity range by at least 3 points on the photosensitivity scale in at least one eye condition (during closure, closed, open) is observed in at least 3 of the 4 patients (with complete suppression in at least 2 patients) in the first cohort, the dose level of JNJ-26489112 may be reduced in subsequent cohorts until the reduction or suppression of photosensitivity is seen in fewer than 2 out of 4 patients in one cohort. Once an effective dose has been reached an additional open-label cohort may be enrolled in which no study drug (JNJ-26489112 or placebo) will be administered to patients. Study drug (i.e., JNJ-26489112 or placebo) will be administered orally as single doses on Days 1 to 3. Placebo will be administered on Days 1 and 3, and a single dose of JNJ-26489112 will be administered on Day 2.

ELIGIBILITY:
Inclusion Criteria:

* Males or postmenopausal/surgically sterile females. Post-menopausal is defined as no menses for the 18 months prior to study start. If menses have ceased within 36 months of the start of this study, then plasma follicle stimulating hormone must be elevated to within a post-menopausal range at study screening
* Pre-menopausal surgically sterilized patients must have a negative beta chorionic gonadotropin pregnancy test at screening and at Day -2
* Women of childbearing potential may be enrolled when results of the reproductive toxicology studies become available, after review of that reproductive toxicology data and upon agreement of the Sponsor and Principal Investigator and the relevant local Ethics Committee, provided these women agree to utilize an acceptable method of birth control
* Body Mass Index (BMI) between 18.5 and 35 kg/m2 (inclusive)
* BMI= weight/height2
* Firm documented diagnosis of idiopathic, photosensitive epilepsy with a generalized photoparoxysmal EEG response
* A photosensitive range in response to intermittent photic stimulation equal to or greater than 4 points in at least one eye condition at screening
* All values for hematology, coagulation, chemistry, and urinalysis within clinically acceptable ranges as they would be for healthy subjects prior to administration of study drug
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Male patients who are not sterile and are unwilling to use condoms for the duration of the study, ensure that their partner practices contraception or refrain from sexual intercourse (and until 90 days after the last dose of study medication).

Exclusion Criteria:

* History of liver or renal insufficiency
* significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic (except epilepsy and febrile seizures), hematologic, psychiatric, or metabolic disturbances.
* Pregnant or lactating female or female insufficiently protected against pregnancy (for female patients of childbearing potential, a negative pregnancy test must be obtained and double-barrier method of contraception must be used starting from screening, throughout the study until follow-up visit), contingent upon satisfactory review of reproductive toxicology study results, and upon agreement of the Principal Investigator, the Sponsor, and the local Ethics Committee).
* Male subjects who are not sterile and are unwilling to use condoms for the duration of the study, ensure that their partner practices contraception or refrain from sexual intercourse (and until 90 days after the last dose of study medication).
* Any serious illness other than epilepsy.
* History of progressive neurological disorder, including brain tumor, active central nervous system infection, demyelinating disease, degenerative or progressive CNS disease.
* Tonic-clonic seizure experienced in the 21-day period prior to Day 1 study drug dose administration (including Day -1).
* Use of herbal medication (including St. John's Wort, garlic extract and herbal teas) or mineral supplements within 14 days prior to study drug administration.
* Use of neuroleptics (typical or atypical) within 60 days prior to study drug administration.
* Use of more than two AEDs, or a change in antiepileptic medication within 30 days prior to study drug administration.
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies (anti-HCV) or Human Immunodeficiency Virus (HIV) antibodies.
* Positive screen for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines). Note: Patients who currently take phenobarbital, mysoline or primidone as antiepileptic therapy and test positive for barbiturates are eligible for study participation. Patients who currently take vigabatrin or frisium as antiepileptic therapy and test positive for benzodiazepines are eligible for study participation.
* Recent history (within previous 6 months) of alcohol or drug abuse.
* Drinks, on average, more than 5 cups of tea/coffee/cocoa/cola per day.
* Smokes on average more than 10 cigarettes per day.
* Clinically significant acute illness within 7 days prior to study drug administration.
* Plasma donation within 7 days prior to study drug administration.
* Legal incapacity or limited legal capacity.
* Likely, in the investigator's opinion, not to cooperate with, or to respect the constraints of the study.
* Donation of 1 or more units (approximately 450 mL) of blood or acute loss of an equivalent amount of blood within 90 days prior to study drug administration.
* Have received an experimental drug or used an experimental medical device within 90 days before the planned start of treatment and/ or plan to use during the planned study participation.
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.
* Patients taking concomitant medications metabolized by CYP2C19 and/or CYP2B6.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The photosensitivity range in each eye condition (during closure, closed, open) based upon the photoparoxysmal electroencepholgram (EEG) response to intermittent photic stimulation (IPS). | Hours 1 to 8 (Day 2) and 25 to 33 postdose (Day 3) with optional assessments at 48, 52, and 56 hours postdose

SECONDARY OUTCOMES:
The safety, tolerability, pharmacokinetics and pharmacokinetic/pharmacodynamic relationship of JNJ-26489112. | Day 1 to Day 3 and an optional Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.